CLINICAL TRIAL: NCT03319875
Title: Evaluation of The Efficacy of Epiduroscopic Discectomy Procedures: A Retroscopic Study
Brief Title: Epiduroscopic Laser Discectomy Procedures
Status: Completed | Type: Observational
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Serbülent Gökhan BEYAZ, Associate Professor, Sakarya University
Other Study IDs: Sakarya University Algology
Record Dates: First submitted 2017-09-26; First posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Disc, Herniated
Keywords: Epiduroscopy; Discectomy; Holmium Yag laser; Lumbar disc herniation; Minimally invasive treatment
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Epiduroscopic Laser Discectomy — Caudal epidural space after passing through sacral hiatus

SUMMARY:
Epiduroscopy or spinal endoscopy is the imaging of the epidural space using a percutaneous and minimally invasive fiberoptic imaging device. The definitive diagnosis and treatment of chronic pain is increasingly prevalent with epiduroscopy. Recently, as a result of these studies it has been reported that laser therapy with epiduroscopy applied discectomy during multiple lesions. Investigators aimed to retrospectively investigate the efficacy of epiduroscopic discectomy procedures performed at the Algology Clinic.

DETAILED DESCRIPTION:
In this study, epiduroscopic discectomy procedures performed between January 2012 and July 2016 at the Algology Clinic of the Department of Anesthesiology and Reanimation, Sakarya University Training and Research Hospital, were examined retrospectively. After approval was received from the Sakarya University Faculty of Medicine's Ethics Committee, patient information was obtained from the KarMed (Kardelen Software, Turkey) hospital information system. Files were scanned from the hospital archive. The age, gender, weight, lumbar disc herniation level, preoperative and postoperative surgical history, amount of physiological saline used during the procedure and duration of the procedure, whether a lumbar epidural steroid (LES) was used during the procedure, the amount of epiduroscopic laser use during the procedure, and complications after the procedure were examined. The Oswestry Disability Index (ODI) and Visual Analogue Scale (VAS) scores were recorded preoperatively, as well as after 2 weeks and 2, 6, and 12 months postoperatively from the patient files.

The 2007 Number Cruncher Statistical System (NCSS, Kaysville, Utah, USA) program was used for statistical analysis. The Student t-test and Mann-Whitney U test were used for descriptive statistical methods (mean, standard deviation, median, frequency, ratio, minimum, maximum) in two groups, as well as the normal distribution of quantitative data. The Kruskal-Wallis test and Mann-Whitney U test were used in the comparison of three groups with no normal distribution. The Pearson Chi-square test was used to evaluate qualitative data, and Spearman's correlation analysis was used to evaluate intervariable relationships. The Friedman and Wilcoxon signed ranks tests were used in the evaluation of three or more follow-up parameters without normal distribution. Diagnostic screening tests (sensitivity, specificity) and receiver operating characteristic (ROC) analysis were used to determine the cutoff value for age. Significance was evaluated at the level of p < (0.01).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with low back and / or leg pain for at least 3 months or more
2. Patients who do not benefit from conservative treatment
3. In patients who underwent Lumbar MRI examinations and had axial sheaths with a herniation of 3 mm or more

Exclusion Criteria:

1. Patients with bleeding diathesis in preoperative laboratory tests
2. Patients with any local or systemic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with low back and / or leg pain attached to the Lomber disc hernia were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2017-06-25 (Actual)

PRIMARY OUTCOMES:
Patients Visual Analog Scale (VAS) scores were assessed retrospectively from hospital information system. Files have been scanned from the hospital archive. | One year
  VAS is a scale that assesses the intensity of pain during rest or activity of the patient. VAS score of 0 indicates no pain and a value of 10 indicates unbearable pain
Oswestry Disability Index (ODI) scores were assessed retrospectively from hospital information system. Files have been scanned from the hospital archive. | One year
  ODI is an evaluation questionnaire that questions how much the pain affects the person's daily activities. It consists of 10 subgroups and each section contains 6 questions. Each episode has 0 points for the first option and 5 points for the sixth option. Subgroups are questioning pain severity, self-care, lifting-carrying, walking, sitting, standing, sleeping, sexual life, travel and social life. As the total score increases, the level of disability also increases.

IPD SHARING:
Plan to Share IPD: No